CLINICAL TRIAL: NCT05961384
Title: A Phase 1, Open-Label Study Of The Absorption, Metabolism, And Excretion Of [14C]-Baxdrostat Following A Single Oral Dose In Healthy Male Subjects
Brief Title: Phase 1 Study to Determine the Metabolism and Clearance of Baxdrostat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN-107-117
Record Dates: First submitted 2023-07-03; First posted 2023-07-27 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
Keywords: pharmacokinetics (PK); metabolism; baxdrostat
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 10 mg [14C]-bexdrostat (Experimental): single oral dose of 10 mg baxdrostat containing 100 μCi of [14C] baxdrostat
  Interventions: Drug: baxdrostat

INTERVENTIONS:
Drug: baxdrostat — a blood pressure lowering drug, oral dose
  Other Names: CIN-107

SUMMARY:
This was a Phase 1, open-label, single dose study in healthy male subjects. The goals of this clinical trial were to determine how baxdrostat might be absorbed and metabolized using radioactive [14C] labeled baxdrostat. Subjects were administered a single oral dose of 10 mg containing approximately 100 μCi of [14C] baxdrostat. Subjects were to be confined to the study site for 9 to 15 days for blood, urine, and feces collections.

ELIGIBILITY:
Subjects must meet the following inclusion criteria:

* Be males of any race between 18 and 55 years of age
* Have a body mass index between 18.0 and 32.0 kg/m2
* Be in good health, determined by no clinically significant findings from medical history
* Have normal renal function, defined as estimated GFR ≥70 mL/min/1.73 m2
* Agree to use contraception
* Be able to comprehend and willing to sign an ICF and to abide by the study restrictions
* Have a history of a minimum of 1 bowel movement per day
* Agree to refrain from donation of sperm from check-in until 90 days after discharge

Main Exclusion Criteria:

* Significant history or clinical manifestation of any diseases as determined by the investigator
* Prolonged QTcF (>450 msec)
* Confirmed (eg, 2 consecutive measurements) systolic BP >140 or <90 mmHg, diastolic BP >90 or <50 mmHg, and pulse rate >100 or <45 beats per minute (bpm).
* Postural tachycardia (ie, >30 bpm upon standing) or orthostatic hypotension (ie, a fall in systolic BP of ≥20 mmHg or diastolic BP of ≥10 mmHg upon standing).
* Serum potassium >upper limit of normal (5.3 mmol/L; ULN) of the reference range and serum sodium <lower limit of normal (135 mmol/L) of the reference range
* Aspartate aminotransferase, alanine aminotransferase, or total bilirubin values >1.2 × ULN.
* A known history of porphyria, myopathy, or active liver disease
* Use of any prescription medications
* Corticosteroid use (systemic or extensive topical use) within 3 months prior to dosing
* Subjects who have participated in more than 3 radiolabeled drug studies in the last 12 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Total radioactivity recovery in urine and feces following administration of [14C] baxdrostat. | 1 to 15 days after dosing
  Measurement of total radioactivity recovery in urine and feces to determine the routes, rates of elimination, and mass balance of total radioactivity from [14C] baxdrostat.
Area under the curve [AUC] of baxdrostat and its primary metabolite (CIN-107M) following administration of [14C] baxdrostat to healthy male subjects. | 1 to 15 days after dosing
  Area under the curve (AUC)0-∞ and AUC0-last will be determined for baxdrostat and CIN-107M in plasma.
Cumulative baxdrostat and CIN-107M excreted in urine and fraction of baxdrostat renally excreted following administration of [14C] baxdrostat to healthy subjects. | 1 to 15 days after dosing
  Determining cumulative amount of baxdrostat and CIN-107M excreted in urine, clearance of baxdrostat and CIN-107M, and fraction of dose excreted renally (baxdrostat only).
Maximum concentration [Cmax] for baxdrostat and CIN-107M in plasma. | 1 to 15 days after dosing
  Cmax will be determined based on measurement of baxdrostat and CIN-107M in plasma.
Time to maximum concentration [Tmax] for baxdrostat and CIN-107M in plasma. | 1 to 15 days after dosing
  Tmax will be determined based on measurement of baxdrostat and CIN-107M in plasma.
Terminal elimination half-life (t1/2) for baxdrostat and CIN-107M in plasma. | 1 to 15 days after dosing
  t1/2 for baxdrostat and CIN-107M in plasma will be determined based on measurement of baxdrostat and CIN-107M in plasma.

SECONDARY OUTCOMES:
Quantitative metabolic profiles of baxdrostat in plasma and excreta. | 1 to 15 days after dosing
  To determine, where possible, the quantitative metabolite profiles in plasma, urine, and feces after [14C]-baxdrostat
Identification of baxdrostat metabolites in plasma and excreta. | 1 to 15 days after dosing
  To determine, where possible, the chemical structure of major metabolites in plasma, urine, and feces after [14C]-baxdrostat
Incidence of treatment emergent adverse events following administration of [14C] baxdrostat. | 1 to 15 days after dosing
  Incidence of adverse events will be used to assess the safety and tolerability of [14C] baxdrostat when administered to healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Siebers, MD Siebers, MD, Principal Investigator — Labcorp Clinical Research Unit, Madison, Wisconsin, USA 53704
Locations (1):
- Labcorp Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-117&attachmentIdentifier=5f19d8f3-3b9c-4b19-bdec-20fa3b299f06&fileName=CIN-107-117_(1).xml&versionIdentifier=